CLINICAL TRIAL: NCT00230347
Title: Dose Escalation Study Evaluating Stereotactic Radiosurgery for Liver Malignancies
Brief Title: Evaluation of Stereotactic Radiosurgery For Liver Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Albert Koong, Stanford University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEP0003; HEP0003; NCT00230347
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Last update posted 2010-04-01 (Estimated); Status verified 2010-03

CONDITIONS: Cholangiocarcinoma; Liver Cancer; Adenocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma; Liver Neoplasms; Adenocarcinoma | interventions — Radiosurgery

INTERVENTIONS:
Procedure: Stereotactic radiosurgery

SUMMARY:
This study is intended to establish the practicality of treating cancer in the liver with precisely administered single fractions of high-energy radiation using a radiosurgical (cross-firing) technique. A second purpose is to establish a safe dose for such therapy. Finally, the efficacy of radiosurgical ablation of liver tumors, in terms of radiographic response, will be measured.

ELIGIBILITY:
Inclusion Criteria:All the following criteria must be met:

* Liver tumors not to exceed 5 cm in diameter. If this size can be increased at all, that would be beneficial as many liver lesions present at a larger size given the lack of symptoms until they are larger and adequate hepatic function with albumin >3.0, total bilirubin <3, INR 1.8. In the case of patients with known or 7 Dose Escalation Study Evaluating Stereotactic Radiosurgery for Liver Malignancies suspected cirrhosis, patients must have creatinine <1.5 and cannot have uncontrolled ascites, encephalopathy, active or recent gastrointestinal bleed (GIB).
* Age > 18 years old
* Histologically confirmed hepatocellular carcinoma (HCC), intrahepatic cholangiocarcinoma (IHCC), or metastatic adenocarcinoma of the breast/colon. Metastatic tumors of other histologic types or sites of origin may be included if the patients have a life expectancy of 6 months or greater. In the case of suspected HCC in patients with known cirrhosis, noninvasive criteria recommended by the European Association for the Study of Liver Diseases may be used. Hypervascular lesions > 2cm with alpha-fetoprotein (AFP) > 400ng/mL or hypervascular lesions >2cm on at least 2 imaging studies.
* Unresectable disease as determined by a surgeon
* Eastern Clinical Oncology Group performance status 0,1 or 2
* No chemotherapy within 1 month of registration
* No prior radiotherapy to the liver or upper abdominal area
* Life expectancy > 6 months
* Patients with IHCC or HCC with distant metastasis are not eligible for this study.
* For colon cancer patients with metastatic tumor of the liver who are not amenable to surgical resection due to the efficacy of removal of simultaneous lung and liver metastasis. Exclusion Criteria:- Children are excluded because HCC, IHCC, and hepatic metastases rarely occur in this age group. Furthermore, treatment requires a great deal of patient cooperation including the ability to lie still for several hours in an isolated room.
* No laboratory personnel will be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2003-10; Primary Completion 2007-01 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Efficacy of radiosurgical ablation of liver tumors, in terms of radiographic response
Practicality of treating cancer in the liver with precisely administered single fractions of high-energy radiation using a radiosurgical (cross-firing) technique
Safe dose for therapy

CONTACTS AND LOCATIONS:
Overall Officials: Albert Koong, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States